CLINICAL TRIAL: NCT00872404
Title: A Phase II Study of CP-751,871 in Patients With Recurrent and/or Metastatic Squamous Head and Neck Carcinoma
Brief Title: A Study of CP-751,871 in Patients With Recurrent Squamous Head and Neck Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2008/02
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Head and Neck Cancer
Keywords: CP-751,871; squamous cell carcinoma; recurrent or metastatic; after 1st line chemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Recurrence; Neoplasm Metastasis | interventions — figitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): CP-751,871 will be administered as an open-label intravenous solution. Patients will remain under clinical observation for one hour post-infusion
  Interventions: Drug: CP-751,871

INTERVENTIONS:
Drug: CP-751,871 — 20mg/kg/3 weeks

SUMMARY:
This is an open-label phase II, multicenter study. Eligible patients will receive CP-751,871 in monotherapy (20 mg/kg IV infusion on Day 1 of 3-week cycles). Tumor check-up will be performed every 6-8 weeks. Treatment will be continued until disease progression or unacceptable toxicities according to the patient or the investigator.

DETAILED DESCRIPTION:
CP-751,871 will be administered as an open-label intravenous solution. All patients will be treated every 3 weeks until disease progression(by RECIST criteria) or unacceptable toxicity death or discontinuation from the study for any other reason.

Since, head and neck tumors are easily accessible for iterative biopsy, this study will offer the opportunity to get tumor biopsies before and after CP-751,871. Our study will allow translational research with biopsies at crucial timing:

(i) at baseline before any treatment, (ii) during the treatment with CP-751,871 (day 1, second cycle two hours after the injection of CP-751,871).

(iii) for patients with stable disease or partial response, a new biopsy will be performed at the time of disease progression to try to understand the mechanisms of tumor resistance.

The baseline samples will allow an investigation of molecular profiles that reflect an inherent inter-patient variability and which will be predictive of response. Although the number of patients included is low, these data may contribute to understand the mechanisms of response and non-response to CP-751,871. Understanding the mechanisms of response to CP-751,871 will help in the rational design of further clinical trials in head and neck cancer using CP-751,871.

The on-treatment samples will help to dynamically monitor the molecular response to CP-751,871.

The study of involved pathways before and after administration of CP-751,871 could be performed using IHC, DNA sequence analysis and RNA expression profiling. Plasma samples could be also stored for further analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent and/or metastatic head and neck squamous cell carcinoma not amenable to curative treatment with surgery and/or chemotherapy and/or radiation.
2. Recurrence must be confirmed by anatomopathology (cytology or biopsy)
3. At least one measurable lesion by MRI or CT-scan.
4. Failed or relapsing after first line chemotherapy including a platinum* or a taxane-based chemotherapy regimen
5. Patients ineligible for chemotherapy could be included in first line
6. ECOG performance status 0 -2, in stable medical condition
7. Patients must have an expected survival of at least 3 months.
8. Paraffin-embedded tumor tissue available for immunohistochemistry
9. Patients must be over 18 years old and must be able to give written informed consent
10. Women of child-bearing age or sexually active female patients with reproductive potential must have a negative pregnancy test (serum or urine within the 7 days prior to enrollment).
11. Patients must have adequate organ function (Hemoglobin ≥ 8 g/100 ml, Neutrophils ≥ 1,000/mm3, Platelets ≥ 75,000/mm3, total bilirubin <1.5 times the upper limit of normal (ULN) for age (except for Gilbert's syndrome patients), serum alanine aminotransferase (ALT) <2.5 ´ ULN for age, aspartate aminotransferase (AST) <2.5 ´ ULN for age , serum creatinine £1.5 x ULN for age
12. Acceptance of giving 20 ml of blood for eventual research at baseline
13. Acceptance of giving two plasma samples (3ml) at baseline and after 3 weeks of treatment
14. Signed informed consent prior to beginning protocol specific procedure
15. Sexually active patients must use effective contraception during the period of therapy and up to 150 days after the last dose of CP-751,871. Acceptable contraception includes, but is not limited to: oral hormone therapy, partner vasectomy, or double barrier contraception (which is defined as a male condom plus spermicide in combination with either a female condom, or diaphragm, or cervical cap or intrauterine device).

Exclusion Criteria:

1. Non-squamous head and neck cancer
2. Nasopharynx cancer
3. Brain metastases
4. More than two lines of chemotherapy for palliative treatment (except if chemotherapy was given as a part of a multimodal treatment given with a curative intent)
5. Surgery or irradiation or investigational drugs within 4 weeks before study inclusion
6. Significant active cardiac disease including: uncontrolled high blood pressure, unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, or serious cardiac arrhythmias
7. Subjects who are receiving chronic high dose immunosuppressive steroid therapy within 2 weeks prior to enrollment (³100 mg prednisone per day or >40 mg dexamethasone per day).
8. Other uncontrolled illnesses (active infections requiring antibiotics, bleeding disorders, uncontrolled diabetes …)
9. Previous malignancy, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
10. Other concomitant anticancer therapies.
11. Previous treatment with anti-EGFR therapy is not an exclusion criteria.
12. Prior anti-IGF-1R therapy
13. Organic brain syndrome or significant psychiatric abnormality that would preclude participation in the full protocol and follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of CP-751,871 alone in patients with head and neck cancer in term of overall response rate and stable disease (RECIST) | 8 weeks

SECONDARY OUTCOMES:
To Determine the safety profile of CP-751,871 alone in patients with head and neck cancer. To Determine the efficacy of CP-751,871 alone in patients with head and neck cancer: progression-free survival and survival | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Machiels, MDPhD, Principal Investigator — Cliniques Universitaires Saint-Luc-UCL
Locations (2):
- Belgium (2):
  - Cliniques universitaires Mont-Godinne, Yvoir, Namur
  - Cliniques Universitaires Saint-Luc, Brussels